CLINICAL TRIAL: NCT03451682
Title: Effects of Procyanidine on Semen Parameters and DNA Fragmentation Index During Cryopreservation of Abnormal Human Semen Samples: a Prospective, Double-blind Trial
Brief Title: Effects of Procyanidine on Semen Parameters and DNA Fragmentation Index During Cryopreservation of Abnormal Human Semen Samples
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aristotle University Of Thessaloniki (Other)
Collaborators: Sohag University (Other)
Responsible Party: Principal Investigator, E.M. Kolibianakis, Associate Professor, Aristotle University Of Thessaloniki
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: UHR-14
Record Dates: First submitted 2018-02-20; First posted 2018-03-02 (Actual); Last update posted 2018-03-02 (Actual); Status verified 2018-02

CONDITIONS: Spermatogenesis and Semen Disorders; DNA Double Strand Break
MeSH Terms: interventions — procyanidin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- procyanidine group (Experimental)
  Interventions: Dietary Supplement: procyanidine
- Control group (No Intervention)

INTERVENTIONS:
Dietary Supplement: procyanidine — Natural antioxidant
  Arms: procyanidine group

SUMMARY:
Cryopreservation is the storage of biological material at subzero temperatures at which biochemical processes of cell metabolism and the biochemical reactions that lead to cell death are slowed, interrupted or stopped.Many investigators have focused on the use of antioxidants in the freezing media to reduce the negative effects of reactive oxygen species(ROS) on spermatozoa and in this context addition of vitamin E to cryoprotective medium enhanced the post-thaw sperm motility and preserved sperm DNA integrity , superoxide dismutase (SOD) and catalase (CAT) were added to boar spermatozoa freezing media and they not only increased sperm motility and viability but also decreased post-thaw ROS generation which led to improvement in results of in vitro fertilizing with thawed spermatozoa.However, the impact of in vitro addition of proanthocyanidins to human semen before cryopreservation on post-thawing semen parameters, DFI has not been studied yet. The research question evaluated in the current study was whether semen samples of infertile men supplemented or not with procyanidine before cryopreservation, differ in post-thawing semen parameters and sperm DNA fragmentation index (DFI).

ELIGIBILITY:
Inclusion Criteria:

Infertility defined as:

* At least twelve (12) months of non-achieving pregnancy despite unprotected sexual intercourse or six (6) months, if the female is > 35 years of age AND
* At least two (2) semen analyses with at least one abnormal parameter (sperm concentration, motility and morphology), according to WHO 2010 criteria.
* Not on any type of infertility treatment for the last three (3) months
* Sperm concentration > 8 x 106/ml and semen volume at least 2.5 ml for technical reasons.
* Normal hormonal profile (TSH, FSH, LH, total testosterone, prolactin)
* Seminal white blood cells < 1 x 106/ml
* No abnormalities in scrotal ultrasound.

Exclusion Criteria:

* Underlying genetic cause of infertility
* History of undescended testis (cryptorchidism)
* History of orchidectomy
* History of testicular cancer
* History of severe cardiac, hepatic or renal disease.
* History of endocrine disease (primary or secondary hypogonadism, hyperprolactinemia, thyroid disease, pituitary or adrenal disease)
* History of epididymo-orchitis, prostatitis, genital trauma, testicular torsion, inguinal or genital surgery
* History of systemic disease or treatment during the last three (3) months
* Positive sperm culture for Chlamydia or Ureaplasma urealyticum
* Female infertility factors
* Body mass index (BMI) > 30 kg/m2
* Participation in another interventional study and a likelihood of being unavailable for follow-up.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2017-08-03 (Actual); Primary Completion 2018-01-10 (Actual); Study Completion 2018-02-05 (Actual)

PRIMARY OUTCOMES:
Progressive sperm motility | 3 Hours after ejaculation and immediately after thawing with or without Procyanidine
  percentage (%) of decrease

SECONDARY OUTCOMES:
Sperm DNA fragmentation index | 3 Hours after ejaculation and immediately after thawing with or without Procyanidine
  percentage (%) of increase
Sperm morphology | 3 Hours after ejaculation and immediately after thawing with or without Procyanidine
  percentage (%) of decrease
Sperm vitality | 3 Hours after ejaculation and immediately after thawing with or without Procyanidine
  percentage (%) of decrease

CONTACTS AND LOCATIONS:
Locations (1):
- Stratis Kolibianakis, Thessaloniki, Greece